CLINICAL TRIAL: NCT04218929
Title: Evaluation of Growth, Safety, and Efficacy of an Infant Formula for Healthy Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ByHeart (Industry)
Collaborators: Paidion Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SS-101-18
Record Dates: First submitted 2019-12-12; First posted 2020-01-06 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Infants; Newborn
Keywords: Infant; Infant Formula; Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Formula (SF) (Experimental): New infant formula for term infants
  Interventions: Other: Study Formula (SF)
- Comparator Formula (CF) (Active Comparator): Commercially available infant formula for term infants
  Interventions: Other: Comparator Formula (CF)
- Human Milk Reference Group (No Intervention): Human milk

INTERVENTIONS:
Other: Study Formula (SF) — New infant formula for term infants fed ad lib
  Arms: Study Formula (SF)
Other: Comparator Formula (CF) — Commercially available infant formula for term infants fed ad lib
  Arms: Comparator Formula (CF)

SUMMARY:
The purpose of this study is to demonstrate that a new infant formula for term infants supports age-appropriate growth. This study is designed in accordance with Good Clinical Practice guidelines and the requirements of the Code of Federal Regulations, 21CFR106.96. In this randomized, controlled trial (RCT), healthy, term, formula-fed (FF) infants will be randomized to one of two infant formulas: a standard, commercially-available infant formula for term infants (CF) or the study formula for term infants (SF) for 16 weeks. A reference group of human milk-fed infants will also be enrolled. The primary efficacy objective is to compare the growth of infants randomized to the study infant formula (SF) versus growth of infants randomized to the standard commercial infant formula (CF).

ELIGIBILITY:
Inclusion Criteria:

* Term (no less than 37 weeks, 0 days and less than 42 weeks, 0 days), singleton infant.
* Birth weight of greater than or equal to 2500 grams.
* Designated healthy by a physician.
* Less than or equal to 14 days of age at enrollment.
* If formula fed, exclusively consuming and tolerating a cow's milk infant formula at enrollment and have a parent who agrees to feed the study formula as a sole source of nutrition for a minimum of 16 weeks.
* If human milk fed, predominantly consuming and tolerating human milk and have a mother/parent who plans to predominantly feed human milk as sole source of nutrition for a minimum of 16 weeks.
* Weight for age greater than or equal to 5th percentile and less than or equal to 95th percentile at enrollment.
* Length for age greater than or equal to 5th percentile and less than or equal to 95th percentile at enrollment.
* Head circumference for age greater than or equal to 5th percentile and less than or equal to 95th percentile at enrollment.
* Weight for length greater than or equal to 5th percentile and less than or equal to 95th percentile at enrollment.
* Not currently receiving and have a parent/guardian who does not plan to give pre- and/or pro-biotics for the full duration of the study.
* Not currently participating in an interventional clinical trial and have a parent(s) or legal guardian(s) who agree not to enroll the infant in an interventional clinical trial while participating in this trial.
* Have parent(s) or legal guardian(s) who are capable of completing the written records, questionnaires, and study procedures required by the protocol.
* Have a parent(s) or legal guardian(s) who have read and voluntarily signed the Institutional Review Board Informed Consent prior to study participation.

Exclusion Criteria:

* Evidence of any anatomic or physiologic condition that would interfere with normal growth, development, or feeding.
* Infants required to take medications know to influence growth and development.
* Maternal history with known adverse effects on the fetus and/or the newborn infants.
* Family history of cow milk protein allergy or soy intolerance/allergy.
* Infants receiving any amount supplemental human milk with infant formula or visa-versa at time of enrollment.
* Infants from a multiple birth.

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Weight Gain Velocity | 0 - 16 weeks
  G/D

SECONDARY OUTCOMES:
Weight Measures | 0 - 16 weeks
  KG
Length Measures | 0 - 16 weeks
  CM
Length Gain Velocity | 0 - 16 weeks
  CM/D
Head Circumference Measures | 0 - 16 weeks
  CM
Weight for age Z-scores | 0 - 16 weeks
  Weight for age Z-scores compared to World Health Organization (WHO) growth standards
Length for age Z-scores | 0 - 16 weeks
  Length for age Z-scores compared to WHO growth standards
Head circumference for age Z-scores | 0 - 16 weeks
  Head circumference for age Z-scores compared to WHO growth standards
Weight for length Z-scores | 0 - 16 weeks
  Weight for length Z-scores compared to WHO growth standards
72-hr record of formula intake at each study visit | 0 - 16 weeks
  OZ/D
Blood concentrations of Interleukin-6 (pg/mL), Interleukin-10 (pg/mL), and tumor necrosis factor-alpha (pg/mL) | 16 weeks
  Concentration
Blood concentrations of amino acids (umol/L) | 16 weeks
  Concentration
Human milk composition (concentrations of proteins, lipids, carbohydrates, vitamins, and minerals | 3 weeks, 7 weeks
  Concentration
Medically-diagnosed adverse events collected throughout the study period | 0 through 16 weeks
  Frequency
Parent rating of infant stool consistency at each study visit | 0 - 16 weeks
  Mean. Quinlan et al Likert scale; 0=no bowel movement, 1=hard [dry hard pellets], 2=formed [definite shape, not dry], 3=soft [no definite shape, pasty], 4=loose [no shape, some water], 5=watery [no shape, mainly water]).
Parent report of infant stool frequency at each study visit | 0 - 16 weeks
  Mean
Parent report of infant disposition (fussiness, crying, gas, spit up, Infant Characteristics Questionnaire) at each study visit | 0 - 16 weeks
  Mean
Stool microbiome | 2 weeks, 16 weeks
  Fecal microbial taxa and community abundance
Stool metabolome | 2 weeks, 16 weeks
  Targeted and Untargeted Metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Devon Kuehn, MD, Study Director — ByHeart, Inc.
Locations (27):
- United States (27):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Watching Over Mothers and Babies, Tucson, Arizona
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - San Gabriel Women's Health, Arcadia, California
  - Northern California Research, Sacramento, California
  - Optum, Colorado Springs, Colorado
  - Topaz Clinical Research, Apopka, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Avanza Medical Research, Pensacola, Florida
  - PAS-Research, Tampa, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Southern Clinical Research, Zachary, Louisiana
  - Sierra Clinical Research, Las Vegas, Nevada
  - Pediatric Associates of Mt. Carmel, Inc, Cincinnati, Ohio
  - Schear Family Practice, Dayton, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Institute of Clinical Research, Mentor, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - Coastal Pediatric Associates, Summerville, South Carolina
  - HMG Primary Care at Sapling Grove, Bristol, Tennessee
  - Jackson Clinic North, Jackson, Tennessee
  - HMG Pediatrics at Kingsport, Kingsport, Tennessee
  - Houston Clinical Research Associates, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - ACRC Trials Plano Pediatrics, Plano, Texas
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuehn D, Zeisel SH, Orenstein DF, German JB, Field CJ, Teerdhala S, Knezevic A, Patil S, Donovan SM, Lonnerdal B. Effects of a Novel High-Quality Protein Infant Formula on Energetic Efficiency and Tolerance: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2022 Oct 1;75(4):521-528. doi: 10.1097/MPG.0000000000003490. Epub 2022 Jun 6. PMID 35666855